CLINICAL TRIAL: NCT05570318
Title: Effect of MiniGo As Add-on to Oral Laxatives for Children with Constipation and Fecal Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Qufora A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: minigo
Record Dates: First submitted 2022-10-05; First posted 2022-10-06 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Functional Constipation; Fecal Incontinence in Children
Keywords: trans anal irrigation; retentive fecal incontinence; low volume TAI
MeSH Terms: interventions — Polyethylene Glycols

STUDY DESIGN:
Intervention Model Description: 50 children randomized into 2 groups. Group a receives current standard treatment, group b receives current standard treatment plus low volume trans anal irrigation as add-on.
Masking Description: Masking not possible, since the add-on treatment requires training of parents and children and is a physical device to be handed out
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Polyethylene glycols (Active Comparator): This group consists of children who have already been treated with oral laxatives (PEG) for at least 2 months, but still experience symptoms of constipation and fecal incontinence.
  Their PEG dosage will be adjusted to the ideal dose for the individual child (this will be evaluated by a health care professional), with the minimum dosage being the maintenance dose of 0,5mg/kg/day, and the maximum dosage being the disimpaction dose of 1,5mg/kg/day
  Interventions: Drug: Polyethylene Glycols
- Polyethylene glycols and low volume trans anal irrigation (Experimental): This group consists of children who have already been treated with oral laxatives (PEG) for at least 2 months, but still experience symptoms of constipation and fecal incontinence. PEG dose will be adjusted in the same manner as in group a, but this group will also receive daily treatment with low volume trans anal irrigation.
  Interventions: Drug: Polyethylene Glycols; Device: Low volume trans anal irrigation

INTERVENTIONS:
Drug: Polyethylene Glycols — To be taken orally on a daily basis throughout the study period (6 weeks) in an adjusted dose.
Device: Low volume trans anal irrigation — To be administered rectally on a daily basis throughout the study period (6 weeks) along with an adjusted dose of polyethylene glycols
  Arms: Polyethylene glycols and low volume trans anal irrigation

SUMMARY:
The goal of this clinical trial is to compare combination therapy with low volume trans anal irrigation (TAI) and oral laxatives to monotherapy with oral laxatives in children with functional constipation and fecal incontinence.

The main questions it aims to answer are:

* Can more efficient treatment be achieved with aforementioned combination therapy?
* Does the well-being of the children change, when they are well treated for their symptoms?
* Is low-volume trans anal irrigation a tolerable treatment method for children?

Participants will be randomized into 2 groups, where one group is treated with current standard treatment of PEG (oral laxatives), and the other group is treated with PEG + daily low volume TAI.

DETAILED DESCRIPTION:
Functional constipation and retentive fecal incontinence is a prevalent health issue in children. The current standard treatment regimen in Denmark consists mainly of behavioral interventions and oral laxative treatment. This treatment leaves a large group of non-responders. Suffering from constipation and fecal incontinence has a negative impact on well-being in children, wherefore treatment of this condition should be improved.

Earlier literature shows that trans anal irrigation (TAI) is an effective means of managing these symptoms, both in children and adults. However, conventional high volume TAI is time consuming (up to 45 minutes-an hour daily) and a cause of discomfort, or even pain. This can lead to low compliance and treatment failure.

Low volume TAI has the potential of bringing about all the positive effects of TAI, but with less time consumption (only few minutes daily) and less discomfort.

In this clinical trial, we will compare how children with functional constipation and fecal incontinence respond to treatment with 1) oral laxatives (PEG) alone versus 2) PEG and low volume TAI with the MiniGo-irrigation system.

The intervention period is 6 weeks, and the treatment takes place at home.

ELIGIBILITY:
Inclusion Criteria:

* age 4-14 years
* medical history with fecal incontinence >1/week on a non-neurogenic but retentive basis (fulfills ROME-IV-criteria)
* non-responsive after min. 2 months treatment with polyethylene glycols and behavioral interventions (set times for toilet use)

Exclusion Criteria:

* Hirschsprungs disease
* anorectal malformations
* use of medications known to cause constipation (eg. anticholinergics)
* former use of low or high volume TAI or enemas

Contraindications for use of MiniGo-irrigation device:

* known stenosis of the rectum or intestinal tract
* colorectal cancer prior to surgical removal
* acute inflammatory bowel disease
* acute diverticulitis
* within 3 months of surgical procedures in the rectum or intestinal tract
* within 4 weeks of endoscopic polypectomy
* ischemic colitis

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Fecal incontinence episodes | 6 weeks
  Seeks to measure if there is any significant difference in the amount of fecal incontinence episodes between the two groups after the study period

SECONDARY OUTCOMES:
Well-being | 6 weeks
  Seeks to measure if the well-being of the children changes when their symptoms are treated. Measured using the WHO-5-well being index
Tolerability of low volume TAI | 6 weeks
  Seeks to investigate whether low volume TAI is tolerated by the children, or if the system causes pain or discomfort.
Constipation symptoms | 6 weeks
  Seeks to investigate whether constipation symptoms (based on ROME-IV criteria) change after treatment

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Aalborg Universitetshospital, Aalborg, Vælg Provins
  - Aarhus Universitetshospital, Aarhus, Vælg Provins
  - Regionshospitalet Gødstrup, Herning, Vælg Provins

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Larsen SO, Axelgaard S, Jonsson IM, Brodersen B, Kristensen SB, Nielsen BR, Hagstrom S, Borch L. Efficacy of low volume transanal irrigation in children with retentive fecal incontinence: A randomized controlled trial. J Pediatr Gastroenterol Nutr. 2026 Feb;82(2):425-433. doi: 10.1002/jpn3.70279. Epub 2025 Nov 18. PMID 41250992